CLINICAL TRIAL: NCT01902628
Title: An Observational, Prospective Study to Evaluate the Hemoglobin Levels in Non-Dialysis Chronic Kidney Disease Subjects With Renal Anemia, Treated With MIRCERA (Methoxy-Polyethylene-Glycol-Epoetin Beta)
Brief Title: OPTIMA: An Observational Study of Mircera (Methoxy Polyethylene Glycol-Epoetin Beta) in Participants With Chronic Kidney Disease Stages 3 and 4 Not on Dialysis
Acronym: OPTIMA
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28261
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with CKD: This single cohort included participants with CKD not receiving dialysis (Stages 3 and 4), with renal anemia, treated with MIRCERA according to usual clinical practice.

SUMMARY:
This prospective observational study evaluated the efficacy and safety of Mircera (methoxy polyethylene glycol-epoetin beta) in chronic kidney disease participants on dialysis with renal anemia. Participants initiated on treatment with Mircera according to the Summary of Product Characteristics and standard clinical practice were followed for 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Participants with chronic kidney disease (CKD) not on dialysis with renal anemia (CKD Stages 3 & 4)
* Initiated on Mircera treatment (participants may have received Mircera treatment for up to 3 months before study enrollment)
* Life expectancy > 10 months

Exclusion Criteria:

* Malignant disease
* Significant or acute bleeding
* Poorly controlled hypertension
* Blood transfusion during the previous 2 months
* Hypersensitivity to Mircera or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic kidney disease (CKD) not on dialysis with renal anemia (CKD Stages 3 & 4) initiated on Mircera therapy
Sampling Method: Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2016-09-04 (Actual); Study Completion 2016-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Greece (24):
  - Uni Hospital of Alexandroupoli; Nephrology Dept., Alexandroupoli
  - Laiko General Hospital; Nephrology Div., Athens
  - Red Cross Hospital;Nephrology Dpt., Athens
  - General Hospital Of Athens G.Gennimatas; Nephrology, Athens
  - Ippokrateion Gen. Hospital Of Athens; 2nd University Clinic Of Internal Medicine, Diabetes Center, Athens
  - Kyanos Stavros Private Hospital; Nephrologic Clinic, Athens
  - General Hospital Of West Attikis; Nephrology, Athens
  - University Hospital Attikon ; Pathology Clinic, Athens
  - Nikea General Hospital; Nephrologic Clinic, Athens
  - General Hospital Of Dramas; Dialysis Center Unit, Drama
  - University Hospital Of Heraklion; Nefrologiki Clinic, Heraklion
  - Uni Hospital of Ioannina; Nephrology Dept., Ioannina
  - General Hospital Of Katerinis; Nephrology Unit, Katerini
  - General Hospital of Kilkis; Nephrology, Kilkis
  - Univeristy Hospital of Larissa; Nephrology, Larissa
  - Agios Andreas General Hospital; Nephrology, Pátrai
  - Olympion Therapeytirion; Nefrology, Pátrai
  - General Hospital Tzanio ; Nephrology, Piraeus
  - General Hospital Of Serres; Nephrology, Serres
  - AXEPA Pathology Section; A Pathology Clinic, Thessaloniki
  - Thermi Private Clinic; Nephrology, Thessaloniki
  - Agios Loukas Private Clinic; Nephrology, Thessaloniki
  - Thessaliki Nossileytiki; Nephrology, Volos
  - General Hospital of Xanthi; Nephrology, Xánthi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With CKD
Started | 437
Completed | 354
Not Completed | 83
Not completed — Withdrawal of participant's consent | 7
Not completed — Adverse Event | 41
Not completed — Lost to Follow-up | 35

BASELINE CHARACTERISTICS:
Arm/Group | Participants With CKD
Number analyzed (Participants) | 437
Age, Continuous [Median (Full Range); unit: years] | 76 [23 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230
  Male | 207

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hemoglobin Levels Within 10.0 - 12.0 g/dL at Months 8-10
Description: g/dL = grams per deciliter
Time Frame: Months 8 to 10
Population: The intent-to-treat population included all eligible participants who received at least one dose of MIRCERA during the observational period, and who had evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With CKD
Number analyzed (Participants) | 437
percentage of participants | 51.2

2. Secondary Outcome: Percentage of Participants With Hemoglobin Levels Within the Following Ranges: 11.0 - 12.0 g/dL, 11.0 - 13.0 g/dL, and 10.0 - 13.0 g/dL at Months 8-10
Description: g/dL = grams per deciliter
Time Frame: Months 8 to 10
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Participants With CKD
Number analyzed (Participants) | 437
percentage of participants
  10.0 - 13.0 g/dL | 68.8
  11.0 - 12.0 g/dL | 35.4
  11.0 - 13.0 g/dL | 53

3. Secondary Outcome: Percentage of Participants With MIRCERA Dose Adjustments
Description: Changes in Mircera dose since last visit are reported. The numbers of participants for which data were not reported are also indicated.
Time Frame: Up to 10 months
Population: The intent-to-treat population included all eligible participants who received at least one dose of MIRCERA during the observational period, and who had evaluable data. Number analyzed indicates number of participants evaluated at specific time points.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With CKD
Number analyzed (Participants) | 437
percentage of participants
  1 Month, Dose Decreased: number analyzed (Participants) | 429
  1 Month, Dose Decreased | 13
  2 Months, Dose Decreased: number analyzed (Participants) | 422
  2 Months, Dose Decreased | 12.4
  3 Months, Dose Decreased: number analyzed (Participants) | 408
  3 Months, Dose Decreased | 10.6
  4 Months, Dose Decreased: number analyzed (Participants) | 399
  4 Months, Dose Decreased | 11
  5 Months, Dose Decreased: number analyzed (Participants) | 388
  5 Months, Dose Decreased | 11.6
  6 Months, Dose Decreased: number analyzed (Participants) | 381
  6 Months, Dose Decreased | 10.2
  7 Months, Dose Decreased: number analyzed (Participants) | 374
  7 Months, Dose Decreased | 10.2
  8 Months, Dose Decreased: number analyzed (Participants) | 366
  8 Months, Dose Decreased | 9.6
  9 Months, Dose Decreased: number analyzed (Participants) | 358
  9 Months, Dose Decreased | 8.2
  10 Months, Dose Decreased: number analyzed (Participants) | 354
  10 Months, Dose Decreased | 8.2
  1 Month, Same Dose: number analyzed (Participants) | 429
  1 Month, Same Dose | 58
  2 Months, Same Dose: number analyzed (Participants) | 422
  2 Months, Same Dose | 54
  3 Months, Same Dose: number analyzed (Participants) | 408
  3 Months, Same Dose | 54.4
  4 Months, Same Dose: number analyzed (Participants) | 399
  4 Months, Same Dose | 50.4
  5 Months, Same Dose: number analyzed (Participants) | 388
  5 Months, Same Dose | 53.8
  6 Months, Same Dose: number analyzed (Participants) | 381
  6 Months, Same Dose | 51
  7 Months, Same Dose: number analyzed (Participants) | 374
  7 Months, Same Dose | 54.6
  8 Months, Same Dose: number analyzed (Participants) | 366
  8 Months, Same Dose | 55.8
  9 Months, Same Dose: number analyzed (Participants) | 358
  9 Months, Same Dose | 60
  10 Months, Same Dose: number analyzed (Participants) | 354
  10 Months, Same Dose | 59.6
  1 Month, Dose Increased: number analyzed (Participants) | 429
  1 Month, Dose Increased | 18.4
  2 Months, Dose Increased: number analyzed (Participants) | 422
  2 Months, Dose Increased | 14.4
  3 Months, Dose Increased: number analyzed (Participants) | 408
  3 Months, Dose Increased | 12.8
  4 Months, Dose Increased: number analyzed (Participants) | 399
  4 Months, Dose Increased | 12.8
  5 Months, Dose Increased: number analyzed (Participants) | 388
  5 Months, Dose Increased | 10.6
  6 Months, Dose Increased: number analyzed (Participants) | 381
  6 Months, Dose Increased | 14.4
  7 Months, Dose Increased: number analyzed (Participants) | 374
  7 Months, Dose Increased | 10.4
  8 Months, Dose Increased: number analyzed (Participants) | 366
  8 Months, Dose Increased | 9.2
  9 Months, Dose Increased: number analyzed (Participants) | 358
  9 Months, Dose Increased | 9.4
  10 Months, Dose Increased: number analyzed (Participants) | 354
  10 Months, Dose Increased | 11.2
  1 Month, Data Not Reported: number analyzed (Participants) | 429
  1 Month, Data Not Reported | 10.4
  2 Months, Data Not Reported: number analyzed (Participants) | 422
  2 Months, Data Not Reported | 19.2
  3 Months, Data Not Reported: number analyzed (Participants) | 408
  3 Months, Data Not Reported | 22.4
  4 Months, Data Not Reported: number analyzed (Participants) | 399
  4 Months, Data Not Reported | 25.8
  5 Months, Data Not Reported: number analyzed (Participants) | 388
  5 Months, Data Not Reported | 24
  6 Months, Data Not Reported: number analyzed (Participants) | 381
  6 Months, Data Not Reported | 24.4
  7 Months, Data Not Reported: number analyzed (Participants) | 374
  7 Months, Data Not Reported | 24.8
  8 Months, Data Not Reported: number analyzed (Participants) | 366
  8 Months, Data Not Reported | 25.4
  9 Months, Data Not Reported: number analyzed (Participants) | 358
  9 Months, Data Not Reported | 22.4
  10 Months, Data Not Reported: number analyzed (Participants) | 354
  10 Months, Data Not Reported | 21

4. Secondary Outcome: Number of Participants With Serious Adverse Events (AEs) and Non-Serious AEs
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug. A serious AE is any experience that suggests a significant hazard, contraindication, side effect, or precaution.
Time Frame: Up to 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With CKD
Number analyzed (Participants) | 437
Participants
  Serious AEs | 56
  Non-Serious AEs | 37

ADVERSE EVENTS:
Time Frame: Up to 10 months
Arm/Group | Participants With CKD
Serious Adverse Events (participants affected / at risk) | 56/437
Other Adverse Events (participants affected / at risk) | 37/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With CKD (N=437)
Anaemia (Blood and lymphatic system disorders) | 6
Leukocytosis (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 1
Cardiorenal syndrome (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death (General disorders) | 3
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Gastroenteritis (Infections and infestations) | 2
H1N1 influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Glomerulosclerosis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Haemodialysis (Surgical and medical procedures) | 1
Peritoneal dialysis (Surgical and medical procedures) | 1
Shock (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With CKD (N=437)
Vertigo (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Catheter site injury (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Chlamydial infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 1
Testicular abscess (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 7
Head injury (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
International normalised ratio increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Haemodialysis (Surgical and medical procedures) | 1
Oral surgery (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Study limitations include the absence of a control group and the observational design of the study. In addition, differences between subgroups found in non-interventional studies cannot be used to infer causality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.